CLINICAL TRIAL: NCT04426552
Title: Dexmedetomidine Versus Sevoflurane Inhalation for Fibreoptic Nasotracheal Intubation in Children With Anticipated Difficult Intubation
Brief Title: Dexmedetomidine Versus Sevoflurane in Children With Anticipated Difficult Intubation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0304285
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Craniofacial Abnormalities; Mandibular Hypoplasia
MeSH Terms: conditions — Craniofacial Abnormalities; Micrognathism | interventions — Dexmedetomidine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): have a bolus of dexmedetomidine one μg/kg (Precedex; Hospira, Inc, Lake Forest, IL) administered for 10 minutes, followed by a continuous infusion at 0.7 μg • kg-1 • h-1 during FOI
  Interventions: Drug: dexmedetomidine
- Sevoflurane (Active Comparator): (sevoflurane) will be preoxygenated using face mask with 100% oxygen for 3 min to increase oxygen reserve and then inhalational induction will be started with sevoflurane in 100% oxygen using Ayre's piece circuit/MapelsonD circuit according to age and weight of the patient while performing fiberoptic intubation
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: dexmedetomidine — will have a bolus of dexmedetomidine one μg/kg (Precedex; Hospira, Inc, Lake Forest, IL) administered for 10 minutes, followed by a continuous infusion at 0.7 μg • kg-1 • h-1 during FOI
  Arms: Dexmedetomidine
Drug: sevoflurane — preoxygenated using face mask with 100% oxygen for 3 min to increase oxygen reserve and then inhalational induction will be started with sevoflurane in 100% oxygen using Ayre's piece circuit/MapelsonD circuit according to age and weight of the patient while performing fiberoptic intubation
  Arms: Sevoflurane

SUMMARY:
difficult problem in the paediatric age group because of their small mouth opening and un-cooperativeness.Currently used methods of sedation for fibreoptic intubation such as benzodiazepines, propofol or opioids may cause respiratory depression, especially when used in high doses

DETAILED DESCRIPTION:
Dexmedetomidine, an a2-agonist, has none-to-minimal respiratory depressant effects, which is clearly a great advantage in handling a critical (unstable, difficult) airway while inducing sedation in both adult and infants. The aim is to compare intubation conditions between dexmedetomidine and sevoflurane inhalation during fibreoptic intubation in pediatric patients with an anticipated difficult intubation

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I and II
* aged 1 year to 3 years
* require general anaesthesia with tracheal intubation for surgical correction of the congenital or acquired pathology that created the difficult airway

Exclusion Criteria:

* parents refusal
* Allergy to drugs

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of intubation | At intubation time
  as assessed by vocal cord movement

CONTACTS AND LOCATIONS:
Overall Officials: Rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab Abd Elraof Abd Elaziz, Alexandria, Smouha, Egypt